CLINICAL TRIAL: NCT04485026
Title: A Randomized Phase II Study of Local Consolidative Radiotherapy Versus Standard of Care Second Line Systemic Therapy in Patients With Oligoprogressive NSCLC on Immune Checkpoint Inhibitors
Brief Title: Local Consolidative Radiotherapy for Oligoprogressive in Non-small Cell Lung Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No enrollments, low patient population as well as a dramatic change in the insurance approval processes for oligoprogressive state with eviCore saying they do not support SBRT in this setting at all.
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00068259; P30CA012197 (NIH); WFBCCC62420 (Other: Wake Forest Baptist Comprehensive Cancer Center)
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Non Small Cell Lung Cancer; Oligoprogressive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Local Consolidative Radiation Therapy Arm (Experimental): Definitive external beam radiation therapy will be delivered to all sites of progressive disease for all patients. The technique used to deliver radiation therapy will be determined by the treating radiation oncologist.
  Interventions: Radiation: Local consolidative radiation therapy
- Standard of Care - Control Arm (Active Comparator): Second line systemic therapy is at the discretion of the treating medical oncologist.
  Interventions: Drug: Standard of care radiation therapy

INTERVENTIONS:
Radiation: Local consolidative radiation therapy — All local consolidative radiation therapy should be delivered using hypofractionated local consolidative radiation therapy (>2 Gy per fraction). Exceptions may be approved on a case by case basis by the trial principal investigator. Three-dimensional conformal radiotherapy (3D-CRT), intensity modulated radiation therapy (IMRT), volumetric modulated arc therapy (VMAT), stereotactic body radiotherapy (SBRT), stereotactic radiosurgery (SRS), and proton beam therapy (PBT) are all acceptable.
  Arms: Local Consolidative Radiation Therapy Arm
Drug: Standard of care radiation therapy — Standard of care palliative radiotherapy to symptomatic lesions is permissible. The dose to symptomatic lesions should not exceed 30 Gy in 10 fractions. Brain metastases will be treated with standard of care CNS therapy throughout the study. This may include (but is not limited to) stereotactic radiosurgery, neurosurgical intervention, whole brain radiotherapy
  Arms: Standard of Care - Control Arm

SUMMARY:
This is a randomized phase II study designed to evaluate the effect of local consolidative radiation therapy (LCT) to all sites of oligoprogressive disease in patients with metastatic non-small cell lung carcinoma who have progressed through first line systemic therapy containing an immune checkpoint inhibitor (ICI).

DETAILED DESCRIPTION:
Primary Objective: To compare overall survival (OS) from the time of the time of randomization between the treatment and control groups.

Secondary Objective(s)

* To compare the extra-CNS PFS2 (EC-PFS2), defined as the time to extracranial disease progression on second line systemic therapy or death from the first day of local consolidative radiation therapy (treatment group) or from the start of second line therapy (control group).
* To evaluate time to initiation of second line systemic therapy or palliative care after completion of local consolidative therapy in the treatment group
* To compare the toxicities in the treatment and control groups;
* To compare overall progression free survival from the time of the first day of local consolidative radiation therapy for the treatment group and from the start of second line therapy for the control group
* To compare the pattern of next progression on second line therapy in the treatment group vs the control group.
* To evaluate local progression in lesions treated with local consolidative radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of non-small cell lung cancer.
* Have completed at least 4 cycles of a first line systemic therapy regimen for metastatic disease that includes a PD-1 axis targeted agent prior to progression. (Patients may be on maintenance/consolidation anti PD-1 axis therapy or have completed maintenance anti PD-1 axis therapy within the last 3 months at the time of progression).
* Initial response of stable disease (SD), partial response (PR) or complete response (CR) in at least one lesion prior to progression as defined by RECIST v1.1 criteria.
* Oligoprogressive disease in 4 or fewer lesions (Progression of the primary tumor and/or regional lymph nodes will be counted as one lesion)
* CNS lesions will not count towards the 4 or fewer progressive lesions if they are all able to be treated with stereotactic radiosurgery.
* Progression by RECIST v1.1 criteria or by PET/CT criteria will be considered progressive disease. Both are not required to determine progressive disease.

Progression for study entry will be defined as by a modified RECIST v1.1 criteria, including: Development of a new lesion; increase in the longest diameter (shortest diameter for lymph node lesions) of any individual lesion by 20% above nadir and a minimal increase of 5 mm.

* In cases of PET/CT, the criteria for progression of PET/CT are: Any individual FDG avid lesion with an uptake greater than twice that of the surrounding tissue on the attenuation corrected image. Any individual FDG avid lesion with greater than 30% increase in 18F-FDG SUV peak, with greater than 0.8 SUV units increase in tumor SUV from the nadir or the pre-enrollment PET/CT in pattern typical of tumor and not of infection/treatment effect per the treating investigator. Visible increase in the extent of 18F-FDG uptake of any lesion by 20% in the longest diameter and an absolute increase of at least 5mm that is not consistent with treatment effect and/or infection per the treating investigator. No more than the following number of progressing lesions in any one organ (including any lesions previously treated with radiation therapy). Less than or equal to four (4) lung lesions (including primary and mediastinal lymph nodes as one lesion). Less than or equal to three (3) liver lesions. Less than or equal to three (3) cumulative vertebral lesions
* At least one non-progressing lesion, which may not have undergone prior definitive local therapy.
* All progressive lesions must be amenable to definitive radiation therapy as determined by the treating radiation oncologist.
* Age of 18 years or greater.
* ECOG Performance Status of 0-2.
* Negative serum or urine pregnancy test within 2 weeks of the date of enrollment
* for women of child-bearing potential.
* Ability to understand and the willingness to sign an IRB-approved informed consent document (either directly or via a legally authorized representative).
* If EGFR and/or ALK status is unknown, the patient is eligible.

Exclusion Criteria:

* Inability to safely treat all progressive lesions with definitive radiation therapy as determined by the treating radiation oncologist
* Patients may not be receiving any other investigational anti-cancer agents.
* Progressive disease in the CNS only.
* Known targetable EGFR mutation or EML4-ALK fusion.
* Progressive cutaneous metastases.
* Progressive disease involving the esophagus, stomach, or intestines.
* Malignant pleural or pericardial effusion at the time of oligoprogression.
* Thoracentesis/thoracoscopic biopsy for a stable or asymptomatic pleural effusion is not required unless the effusion is hypermetabolic on PET/CT or if there are active pleural based metastatic lesions at the time of oligoprogression.
* Effusions that are too small for thoracentesis/pericardiocentesis are considered resolved for the purposes of trial eligibility.
* Pregnant women are excluded from this study because radiation therapy has known potential for teratogenic or abortifacient effects.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements as determined by the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-05-09 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  In each arm overall survival will be defined as the time from randomization to death from any cause. . Patients who are alive at the last follow up at the end of the study will be censored at the date of the last follow up appointment. A comparison of overall survival between the two groups will be made first using bivariate Kaplan-Meier method and then a multivariable Cox proportional hazards model. Participants who do not die during the course of observation will be right censored. Key covariates to be included in multivariable modeling include age, ECOG status, number of progressive treated sites (1 vs 2-4), and PD-L1 status (>=50%; 1%-49%; < 1%).

SECONDARY OUTCOMES:
Time to Progression Between Both Arms | 3 years
  Investigators will compare progression after second line of therapy between both arms first using the bivariate Kaplan-Meier method and then a multivariable Cox proportional hazards model age, ECOG status, number of progressive treated sites (1 vs 2-4), and PD-L1 status (>=50%; 1%-49%; < 1%). RECIST version 1.1 criteria will be used to assess for progression.
Time to Second Line of Systemic Therapy or Palliative Care (Local Consolidative Radiation Therapy Arm Only) | Up to 2 years after the completion of intervention
  The time to the second line systemic therapy or palliative care will be defined as the time from the completion of local consolidation therapy to the first day of cycle 1 of a systemic therapy the patient has not yet received OR the date of hospice enrollment, whichever is sooner. Patients experiencing neither of these events will be censored at last follow up visit. Estimated median time to second line therapy (or palliative care) and corresponding 95% confidence interval as well as estimated proportion (and corresponding 95% confidence interval) of the treatment group who have started second-line therapy (or palliative care) by key time points including 6 months, 1 year, and 2 years after the end of local consolidative therapy.
Incidences of Toxicities | Up to 3 years
  Toxicities will be evaluated per Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Toxicities between the two arms by comparing the proportions with grade 2 or higher, and grade 3 or higher, toxicities of any type at 3, 6, 12, 24 and 36 months following randomization using a chi-square test on the relevant 2x2 contingency table.
Progression Free Survival | Up to 5 years
  Progression free survival will be assessed by a modified RECIST version 1.1 criteria. If any individual target lesion meets RECIST v1.1 criteria - specifically an increase in the longest diameter (shortest diameter for lymph node lesions) of at least 20% and 5 mm absolute increase, the patient will be considered to have progression of disease. The criteria for determining pseudoprogression versus true progression and for mild progression while systemic therapy is held for the delivery of local consolidative radiation therapy in the treatment arm will be used for this outcome measure as well. Repeat oligoprogression will also be counted as progressive disease.
Time to Next Progression Following Local Consolidative Radiation Therapy or Second Line Systemic Therapy | Up to 3 years
  The pattern of next progression following local consolidation therapy (in treatment group) or second line systemic therapy (in control group) into one of three possible mutually exclusive and exhaustive categories: No progression, repeat oligoprogression or polyprogression, and will compare these patterns between the two groups using a chi-square analysis on the resulting 2x3 contingency table.
Proportion of Local of Lesions Treated with Local Consolidative Radiation Therapy That Progress | Up to 5 years
  Investigators will estimate proportion of lesions treated with local consolidative radiation therapy that experienced local progression (yes/no by study end) and construct a 95% confidence interval around this estimate.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farris, MD, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No